CLINICAL TRIAL: NCT03684395
Title: Association Between Socioeconomic Factors and Use of Direct Oral Anticoagulants Versus Standard of Care (Warfarin) in Patients With Non-valvular Atrial Fibrillation in Sweden
Brief Title: Accessibility to New Drugs Versus SOC in Sweden
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18984
Record Dates: First submitted 2018-09-14; First posted 2018-09-25 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Anticoagulation
MeSH Terms: interventions — Dabigatran; apixaban; Standard of Care; Warfarin

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DOACs (Direct Oral Anticoagulants)
  Interventions: Drug: DOACs: Rivaroxaban, Dabigatran, Apixaban
- Standard of care
  Interventions: Drug: Standard of care (Warfarin)

INTERVENTIONS:
Drug: DOACs: Rivaroxaban, Dabigatran, Apixaban — Routinely collected clinical data (secondary data from patients with non-valvular atrial fibrillation in Sweden); no primary data collection
  Groups: DOACs (Direct Oral Anticoagulants)
Drug: Standard of care (Warfarin) — Routinely collected clinical data (secondary data from patients with non-valvular atrial fibrillation in Sweden); no primary data collection
  Groups: Standard of care

SUMMARY:
The healthcare system in Sweden is publicly funded and aims to provide equal access to care irrespective of socioeconomic status. This includes ensuring equity in drug treatment. Socioeconomic disparities have been shown to influence patient management and health outcomes in certain Swedish populations. The Swedish Board of Health and Welfare has stated that the prescription of new drugs, which are more expensive than generic standard of care drugs, might be influenced by patients' socioeconomic status.

To evaluate the association between socioeconomic factors and use of a DOAC (rivaroxaban, dabigatran, or apixaban) or standard of care (warfarin) in patients with NVAF in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years in Sweden with a diagnosis of NVAF (identified using International Classification of Diseases, version 10 [ICD-10]) codes in the National Patient Register) between 1 December 2011 and 31 December 2014 and with a first dispensed prescription for either a DOAC or warfarin following their NVAF diagnosis.

Exclusion Criteria:

* Patients with a dispensed prescription for a DOAC or warfarin prior to the index date (the date of first DOAC/warfarin purchase designated the index date)
* Patients with a dispensed prescription for more than one anticoagulant at index date.
* Patients with valvular atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 68056 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Correlation between socioeconomic factors and use of DOACs vs. Warfarin (as identified from the LISA database before the index date) | approximately 3 years
  Between 1 December 2011 and 31 December 2014;
  Socioeconomic factors:
  * Occupation
  * Education
  * Income
  * Family status
  * Immigrant status

SECONDARY OUTCOMES:
Secular trends in the correlation between socioeconomic factors and use of DOACs (vs. warfarin) - Trends based on the date of prescription by year | approximately 3 years
  Between 1 December 2011 and 31 December 2014; Relationship between socioeconomic factors and access to newly marketed drugs (DOACs as one class which includes Rivaroxaban, Dabigatran and Apixaban) versus standard of care (warfarin) for different calender period.

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm, Sweden